CLINICAL TRIAL: NCT04772261
Title: 13C-Spirulina Breath Test (13C-GEBT) Lot-to-Lot and Biological Variability Study
Brief Title: GEBT Lot-to-Lot and Biological Variability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairn Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO-CD-050
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Gastroparesis
Keywords: Gastroenterology; Gastric emptying breath test
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Lot-to-Lot Variability (Experimental): Participants will be administered up to six different 13C-Spirulina test meal lots
  Interventions: Diagnostic Test: 13C-Spirulina GEBT
- Biological Variability (Experimental): Participants will be administered the same 13C-Spirulina test meal lot on two different occasions
  Interventions: Diagnostic Test: 13C-Spirulina GEBT

INTERVENTIONS:
Diagnostic Test: 13C-Spirulina GEBT — Various lots of 13C-Spirulina GEBT test meals

SUMMARY:
The purpose of this study is to collect information regarding lot-to-lot variability in 13C-Spirulina test meal lets and within-subject biological variability.

DETAILED DESCRIPTION:
In this study participants will participate in one or two arms of the study. In one arm the participants will be administered GEBT tests that contain different 13C-Spirulina/Egg mix drug lots. In the second arm, the participants will be administered GEBT tests from the same 13C-Spirulina/Egg mix drug lot. All GEBT kit lots will be administered according to the FDA-approved labeling.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18-85 years old at time of signing the informed consent form
* Ability to eat test meal and provide breath samples

Exclusion Criteria:

* History or physical exam suggestive of systemic disease such as diabetes mellitus or pathophysiologic disorders such as renal failure, chronic heart disease, chronic respiratory disease, liver disease, or malabsorption.
* History of abdominal surgery except appendectomy
* Use of any medications that may alter gastric motility within two days of the study
* Use of narcotics or anticholinergics within two days of the study
* Females on hormone replacement therapy other than birth control medications
* Pregnancy
* Intolerance or allergy to any component of GEBT test meal
* History of neurologic or psychiatric disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Lot to Lot Variability | up to 3 months
  Participant kPCD values at each measured timepoint from each lot of 13C-Spirulina GEBT test meal will be plotted to compare in vivo results across each lot of material
Lot to Lot Variability | up to 3 months
  Pooled kPCD and standard deviations for each measured timepoint from each lot of 13C-Spirulina GEBT test meal will be calculated and compared for the lot-to-lot comparisons
Lot to Lot Variability | up to 3 months
  Each set of pooled 13C-Spirulina test meal lot kPCD values will be calculated using a t-test or ANOVA to determine statistical equivalence
Biological Variability | Up to 3 months
  Participant kPCD values at each measured timepoint from the same 13C-Spirulina GEBT test meal will be plotted to compare against each other
Biological Variability | Up to 3 months
  Pooled, within subject standard deviations of duplicate measurements of kPCD values at each measured timepoint from the same lot of 13C-Spirulina GEBT test meal will be calculated for biological variation using Bartlett's test for homogeneity of variances

CONTACTS AND LOCATIONS:
Overall Officials: Alex Ryder, MD, PhD, Principal Investigator — Cairn Diagnostics
Locations (1):
- Cairn Diagnostics, Brentwood, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT04772261/Prot_SAP_000.pdf